CLINICAL TRIAL: NCT06118762
Title: A Single-arm, Open, Multicenter Clinical Study of Fruquintinib Combined With Raltitrexed in the Treatment of Metastatic Colorectal Cancer
Brief Title: Clinical Study of Fruquintinib Combined With Raltitrexed in the Treatment of Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-E1-C002
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; Fruquintinib; Raltitrexed
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; raltitrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib combined with Raltitrexed group (Experimental): Fruquintinib combined with Raltitrexed therapy
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib capsule is taken orally once a day, 5 mg each time, and taken for 2 weeks and stopped for 1 week, every 21 days (3 weeks) for a cycle. Raltitrexed: 3 mg/m2 intravenously, on the first day of each cycle, for a treatment cycle of 3 weeks. Combination treatment until toxicity becomes intolerable, disease progression, or death.
  Other Names: Raltitrexed

SUMMARY:
To evaluate the efficacy and safety of Fruquintinib combined with Raltitrexed in the treatment of metastatic colorectal cancer that progressed or could not be tolerated after previous fluorouracil, oxaliplatin, and irinotecan based therapy

DETAILED DESCRIPTION:
To evaluate the progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), overall survival (OS), and safety of Fruquintinib combined with Raltitrexed in 30 patients with metastatic colorectal cancer who had progressed or could not tolerate fluorouracil, oxaliplatin, and irinotecan based therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Age ≥18 years old, gender unlimited;
3. Advanced metastatic colorectal adenocarcinoma confirmed by histopathology;
4. The patient progressed or was intolerant after receiving at least previous standard therapy containing fluorouracil, oxaliplatin, and irinotecan.

   * Each first-line treatment must include one or more chemotherapeutic agents for a duration of ≥1 cycle;
   * Allow pre-adjuvant/neoadjuvant therapy. If recurrence or metastasis occurs during or within 6 months after completion of adjuvant/neoadjuvant therapy, adjuvant/neoadjuvant therapy is considered a failure of first-line chemotherapy for advanced disease;
   * Prior chemotherapy combined with cetuximab or bevacizumab is permitted;
5. Have at least one measurable lesion (RECIST 1.1 standard);
6. Eastern Cooperative Oncology Group (ECOG) physical condition 0-1 score;
7. Expected survival ≥12 weeks;
8. The functions of vital organs during the first 14 days of enrollment meet the following requirements (the use of any blood components and cell growth factors during the first 14 days of enrollment is not allowed) :

   * Absolute neutrophil count ≥1.5×109/L;
   * Platelet ≥80×109/L;
   * Hemoglobin ≥8g/dL;
   * Total bilirubin < 1.5 × upper limit of normal（ULN）;
   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 2.5 × ULN (< 5 × ULN in patients with liver metastasis);
   * Serum creatinine ≤1 × ULN;
   * endogenous creatinine clearance > 50ml/min;
9. Women of childbearing age or men whose partners wish to have children need to take effective contraceptive measures.

Exclusion Criteria:

1. Previous treatment with Fruquintinib or other anti-vascular endothelial growth factor receptor (VEGFR) inhibitors such as Apatinib, Regorafenib, and Anlotinib;
2. Previous treatment with Raltitrexed;
3. Participated in other drug clinical trials and received at least one drug therapy within four weeks prior to enrollment or received other systemic anti-tumor therapy, including chemotherapy, signal transduction inhibitors, hormone therapy, and immunotherapy within four weeks prior to enrollment;
4. The patient currently has a disease or condition that affects drug absorption, or the patient cannot take Fruquintinib orally;
5. The patient currently has gastrointestinal diseases such as gastric and duodenal active ulcers, ulcerative colitis, or active bleeding from unresectable tumors, or other conditions determined by researchers that may cause gastrointestinal bleeding or perforation;
6. Patients with active bleeding or bleeding tendency;
7. History of severe cardiovascular and cerebrovascular diseases:

   * Cerebrovascular accident (excluding lacunar infarction, minor cerebral ischemia, or transient ischemic attack), myocardial infarction, unstable angina, and poorly controlled arrhythmias (including QTc interval ≥ 450ms for men and 470 ms for women) within 6 months prior to first administration of the study drug (QTc interval Fridericia) Formula calculation);
   * New York Heart Association (NYHA) Heart Function Rating > Grade II or left ventricular ejection fraction (LVEF) < 50%;
8. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
9. Clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or C (hepatitis B virus infection regardless of drug control, hepatitis B virus DNA≥1×104 copies /mL or > 2000 IU/ml);
10. There is known to be symptomatic central nervous system metastasis and/or cancerous meningitis. Participants with previously treated brain metastases may participate in the trial if their condition is stable (no evidence of radiographic progression at least 4 weeks prior to initial administration of the trial treatment), repeated radiographic studies confirm no evidence of new brain metastases or enlargement of the original brain metastases, and no steroid therapy is required at least 14 days prior to initial administration of the trial treatment. This exception does not include cancerous meningitis, which should be excluded regardless of whether it is clinically stable;
11. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
12. The patient currently has hypertension that cannot be controlled by drugs, which is prescribed as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after taking antihypertensive drugs;
13. Urine routine indicates urinary protein ≥2+, or 24-hour urinary protein volume > 1.0g;
14. The patients considered by the investigators to be unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death
  The time from enrollment to disease progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 1 year
  Proportion of patients with complete or partial response
Disease control rate (DCR) | through study completion, an average of 1 year
  Proportion of patients assessed as having a complete response, partial response, or stable disease
Overall survival (OS) | Through study completion, an average of 1year
  Patients were enrolled until their death from any cause
Security | Through study completion, an average of 1year
  Safety was evaluated by adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Peng, Director, Study Chair — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China